CLINICAL TRIAL: NCT00516841
Title: A Phase 2, Single-Arm Study of Volociximab Monotherapy in Subjects With Platinum-Resistant Advanced Epithelial Ovarian Cancer or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision to terminate recruitment based on lack of efficacy
Sponsor: Facet Biotech (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206OC201
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer; Peritoneal Neoplasms
Keywords: epithelial ovarian cancer; peritoneal cancer; platinum-resistant ovarian cancer; Platinum-Resistant Advanced Epithelial Ovarian Cancer or Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Carcinoma, Ovarian Epithelial | interventions — volociximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- volociximab (Experimental): 15 mg/kg volociximab once weekly
  Interventions: Drug: Volociximab

INTERVENTIONS:
Drug: Volociximab — 15 mg/kg weekly, IV infusions, for 8 weeks or until disease progression or unacceptable toxicity develops
  Other Names: M200

SUMMARY:
To evaluate the efficacy of voloxicimab when administered at 15 mg/kg qwk in subjects with platinum-resistant, advanced epithelial ovarian cancer or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law (e.g., Protected Health Information [PHI]).
* Females aged ≥18 years old at the time of informed consent.
* Advanced (Stage III or IV), histologically-documented epithelial ovarian cancer or primary peritoneal cancer (excluding small, round-cell histologies).
* Radiologically-documented evidence of progressive disease.
* Platinum-resistant disease defined as having a best response of SD or disease progression during or within 6 months of discontinuing a platinum-based chemotherapy (carboplatinum, cisplatinum, or another organoplatinum compound).
* Progression during or following treatment with topotecan or liposomal doxorubicin.
* Three or fewer prior chemotherapy regimens (including a platinum-based therapy).
* At least 1 measurable target lesion in accordance with RECIST criteria to assess clinical response (tumors within a previously irradiated field are designated as non-target).
* ECOG Performance Status ≤1.
* Life expectancy >12 weeks.
* Available paraffin block or unstained paraffin sections on glass slides containing representative tumor tissue from the most recent tumor biopsy/resection.
* Subjects of child-bearing potential must be willing to practice effective contraception during the study and be willing and able to continue contraception for at least 6 months after their last dose of study treatment (about 5 half lives).

Exclusion Criteria:

* Screening clinical laboratory values:

  * Absolute neutrophil count <1500/µL
  * Platelet count <75,000/µL
  * Hemoglobin <8.5 g/dL (hemoglobin may be supported by transfusion, erythropoietin, or other approved hematopoietic growth factors; darbopoeitin [Aranesp®] is permitted)
  * Serum bilirubin >2.0 x upper limit of normal (ULN)
  * AST and ALT >2.5 x ULN (AST and ALT >5 × ULN for subjects with liver metastasis)
  * Serum creatinine >2.0 mg/dL
  * International normalized ratio (INR) >1.5
  * Activated partial thromboplastin time (aPTT) >1.5 × ULN
* Clinically significant peripheral vascular disease.
* Non-epithelial ovarian tumors.
* Active infection requiring systemic antibiotics, antivirals, or antifungals including HIV/AIDS, hepatitis B, or hepatitis C infection.
* History of abdominal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to Day 1.
* Serious, non-healing wound, or bone fracture.
* Known central nervous system or brain metastases.
* History of uncontrolled psychiatric condition within 6 months prior to Day 1.
* History of other malignancies within 3 years of Day 1, except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of breast, or basal or squamous cell skin cancer.
* Evidence of autoimmune disease including, but not limited to, ulcerative colitis, Crohn's disease, rheumatoid arthritis (RA), systemic lupus erythematosus (SLE) sceloderma, or another diseases in which immune function or immune competence is known to be impaired.
* Any history of lymphoproliferative disorder.
* Known human anti-murine antibody (HAMA) and/or human anti-chimeric antibody (HACA).
* Any medical condition that may be exacerbated by bleeding, including a known bleeding disorder such as a coagulation defect, thrombocytopenia, active gastric or duodenal ulcer, or history of GI bleeding.
* Significant hemoptysis within one year prior to Study Day 1.
* Any investigational, anti-cancer therapy within 6 weeks prior to Day 1.
* Any non-investigational, anti-cancer therapy within 4 weeks prior to Day 1.
* Prior treatment with anti-angiogenic agents.
* Subjects who require treatment with an anti-coagulant with the exception of low-dose Aspirin® (≤81 mg/day), warfarin (≤1 mg/day), or heparin for IV catheter patency.
* Subjects who are taking concomitant immunomodulatory agents including, but not limited to, interferons, interleukins, systemic steroids, cyclosporine, tacrolimus, calcineurin inhibitors, chronic low-dose methotrexate, or azathioprine. (The use of inhaled or intranasal steroids or oral steroids at a dose of ≤10 mg/day prednisone or its equivalent are permitted.)
* Active, unstable severe cardiovascular disease, including poorly controlled angina, congestive heart failure (CHF), arrhythmias, myocardial infarction (MI), cardiomyopathy, atrioventricular (AV) block, electrocardiogram (ECG) evidence of acute ischemia, or significant conduction abnormality.
* History of thromboembolic or cerebrovascular events, such as stroke, or transient ischemic attack (TIA). (Note: Prior history of deep vein thrombosis will not exclude subjects from participating in this study.)
* Pregnant (positive pregnancy test) or lactating.
* Inability to comply with study and follow-up procedures.
* Any condition that, in the opinion of the Investigator, makes the subject unsuitable for study participation.
* Known hypersensitivity to murine or chimeric antibodies.
* Major surgery within 4 weeks prior to Day 1.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by objective response rate (ORR). Tumor response based on RECIST criteria. | Baseline, and every 8 weeks on study

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Matthews, MD, Principal Investigator — Mary Crowley Medical Research Center; Minal Barve, MD, Principal Investigator — Texas Oncology PA, Presbyterian; James Burke, MD, Principal Investigator — Billings Clinic (MCMRC network); Dana Glenn, MD, Principal Investigator — Sharp Hospital; Russell Schilder, MD, Principal Investigator — Fox Chase Cancer Center; Nikki Spellman, MD, Principal Investigator — Indiana University; Michael Gold, MD, Principal Investigator — Oklahoma University Health Science Center; Richard Penson, MD, Principal Investigator — Massachusetts General Hospital; Mark Einstein, MD, Principal Investigator — Montefiore Medical Center; Robert Holloway, MD, Principal Investigator — Florida Hospital Cancer Institute; Deborah Armstrong, MD, Principal Investigator — Johns Hopkins Kimmel Cancer Center; Snehel Bhoola, MD, Principal Investigator — Memorial Health University Medical Center; Eric Winquist, MD, Principal Investigator — London Health Sciences Center; Ernst Lengyel, MD, Principal Investigator — University of Chicago; John Glaspy, MD, Principal Investigator — UCLA JCCC Clinical Research Unit; Krish Tewari, MD, Principal Investigator — UCI Medical Center; C. William Helm, MD, Principal Investigator — James Graham Brown Cancer Center; John Glaspy, MD, Principal Investigator — University of California, Los Angeles; Michael Sawyer, MD, Principal Investigator — Cross Cancer Institute
Locations (23):
- United States (19):
  - UCLA JCCC Clinical Research Unit, Los Angeles, California
  - UCI Medical Center, Orange, California
  - Sharp Hospital, San Diego, California
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Billings Clinic (MCMRC network), Billings, Montana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology PA, Presbyterian, Dallas, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
- Canada (4):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - London Health Sciences Center, London, Ontario
  - McGill University Hospital, Montreal, Quebec